CLINICAL TRIAL: NCT03498079
Title: Prevalence of Mullerian Anomalies and PCO in Egyptian Women
Brief Title: Prevalence of Mullerian Anomalies in Infertile Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Kasr El Aini Hospital (Other); National Research Centre, Egypt (Other); misr Infertility centre ,Alaqsor (Unknown)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Assistant Researcher , National Research centre and Specialist of Obstetrics and Gynecology in Aljazeerah hospital, Aljazeera Hospital
Other Study IDs: mullerian anomalies
Record Dates: First submitted 2018-04-07; First posted 2018-04-13 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Mullerian Anomaly of Uterus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 3D ultrasound — 3D ultrasound will be done to females complaining from primary infertility with mullerian anomalies

SUMMARY:
* Mullerian anomalies are congenital structural anomalies in the uterus .
* Its prevalence is not uncommon .

DETAILED DESCRIPTION:
* PCO is very common in gynecological practice
* Women with mullerian anomalies should be properly evaluated for other gynecological and urological problems

ELIGIBILITY:
Inclusion Criteria:

* females with age between 20-42 years with primary infertility

Exclusion Criteria:

* females with age above 42 years or below 20 years females with secondary infertility

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — females with primary infertility
Study Population: - females with age between 20-42 years with primary infertility
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-04-20 (Estimated); Study Completion 2019-04-25 (Estimated)

PRIMARY OUTCOMES:
the number of participants who will prove to have PCO | within 4 weeks
  diagnosis of PCO by US and by FSH and LH levels

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
we will publish the results which will be obtained from this study